CLINICAL TRIAL: NCT01322386
Title: The Human Gastrointestinal Tract Microbiota in the Setting of Treating Primary Sclerosing Cholangitis and Biliary Atresia With Vancomycin.
Brief Title: Gastrointestinal Microbiota in Primary Sclerosing Cholangitis and Biliary Atresia With Vancomycin
Acronym: PSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kenneth L. Cox, Professor of Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4751
Record Dates: First submitted 2011-02-10; First posted 2011-03-24 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Primary Sclerosing Cholangitis; Biliary Atresia
Keywords: PSC; BA
MeSH Terms: conditions — Cholangitis, Sclerosing; Biliary Atresia | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Vancomycin (Experimental): Vancocin
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Oral 50mg/Kg per day up to maximum of 1500 mg a day for three months.
  Other Names: Vancocin

SUMMARY:
The goals of the proposed work are two fold:

Firstly, to see if the antibiotic vancomycin may be used for the early treatment of Biliary Atresia (BA) and Primary Sclerosing Cholangitis (PSC). The investigators hope to learn what effect Vancomycin has on the bacteria that are present in stool, body fluid or intestinal tissue on someone who has BA and PSC and if so by what mechanism. Secondly, the investigators hope to learn to characterize human intestinal microbial communities (microbiome: the collection or collectivity of microorganisms) using molecular methods, examine the mechanisms of interaction between host and microbiome using genomic approaches, and determine how the microbiome both preserves local health and promotes pathology. The investigators will focus on primary sclerosing cholangitis, biliary atresia, as well as states of health. The composition of the associated microbiome will be assessed based on ribosomal DNA and RNA sequences, and attention will be given to richness (diversity), evenness (relative abundance), and variation with respect to time, person, and anatomic niche. Host response at the adjacent mucosal surface will be assessed based on genome-wide gene expression patterns.

DETAILED DESCRIPTION:
As many as 55 subjects (35 with BA or PSC and 20 Controls) will be involved. We are also recruiting 20 adult patients with either BA, or PSC. The patients will be recruited from Lucile Children's Hospital, Stanford Medical Center, and Stanford Redwood City Campus such as patients with primary sclerosing cholangitis, biliary atresia or other intestinal disorders for whom upper or lower endoscopy is indicated for routine medical management. There may be some participants who are over 18 years of age although the vast majority will be under 18. Vancomycin therapy will be administered to the BA patients (4 weeks)and PSC patients. The PSC patient blood tests would now be done at various intervals: before starting the Vancomycin; every month until their Liver Function Tests are normalized; after their Liver Function Tests are normalized; before stopping the Vancomycin and after they are off the Vancomycin at month 1,3,6,12,and 24. Fecal samples will be taken.

In addition, patients who will already be undergoing either upper or lower intestinal endoscopy for routine diagnostic or therapeutic purposes will be asked to agree to endoscopic mucosal brushings in addition to mucosal biopsies. Some will be patients with a diagnosis of primary sclerosing cholangitis, biliary atresia, or other intestinal disorders for whom upper or lower endoscopy is indicated for routine medical management. Others will have lower intestinal findings (polyps) or complaints (e.g. occult blood in stool), or upper intestinal findings (dyspepsia, reflux), and will be undergoing lower endoscopy (colonoscopy) or upper endoscopy for routine medical management. Up to 2 biopsies will be obtained from the gastric mucosa and of as many as 6 intestinal sites from each patient. In addition the following brushings will be taken: 2 from mid-esophagus, 2 from lesser curvature of the stomach, 2 from the second portion of the duodenum near the ampulla. 2 from the jejunum 5 cm from the Ligament of Trietz, and 2 from the ileum 10 cm from the ileocecal valve. We will also obtain brushing from the tongue. A sample of saliva will be taken.

Fecal specimens will also be collected just prior to bowel preparation for endoscopy/colonoscopy. If the BA patient is already having a Kasai portoenterostomy, done to remove the diseased bile ducts, we would like to take a biopsy of the bile duct. If the patient has a liver biopsy clinically done we would like to keep a 2mm section of it. If the patient has an intraoperative cholangiogram to evaluate the bile ducts we will collect 2.5 cc. of bile fluid. With regards to the controls, who have other intestinal disorders and are also having clinical endoscopies done, we would request a midesophagus biopsy; a biopsy from the antrum and 2 biopsies from the 4th portion of the duodenum. Cell brushings will be taken from the following areas: 2 from mid-esophagus, 2 from lesser curvature of the stomach, 2 from the second portion of the duodenum near the ampulla. 2 from the jejunum 5 cm from the Ligament of Trietz, and 2 from the ileum 10 cm from the ileocecal valve. We will also obtain brushing from the tongue. A sample of saliva will be taken. If the patient is having a colonoscopy done as part of their clinical care we would request a biopsy from the ileum, cecum, and transverse descending rectum. We would also ask for a saliva sample.

The blood tests would now be done at various intervals: before starting the Vancomycin; every month until their Liver Funtion Tests are normalized; after their Liver Function Tests are normalized; before stopping the Vancomycin and after they are off the Vancomycin at month 1,3,6,12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of biliary atresia or primary sclerosing cholangitis.
* Clinical controls who are undergoing upper endoscopy or colonoscopy and do not have biliary atresia or primary sclerosing cholangitis.
* Subjects who have been on oral vancomycin for 1 year for biliary atresia or -

Exclusion Criteria:

* Patients that have taken antibiotics within the last 3 month will be excluded as this will alter the original bacterial flora.

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Cox, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali AH, Damman J, Shah SB, Davies Y, Hurwitz M, Stephen M, Lemos LM, Carey EJ, Lindor KD, Buness CW, Alrabadi L, Berquist WE, Cox KL. Open-label prospective therapeutic clinical trials: oral vancomycin in children and adults with primary sclerosing cholangitis. Scand J Gastroenterol. 2020 Aug;55(8):941-950. doi: 10.1080/00365521.2020.1787501. Epub 2020 Jul 7. PMID 32633158
- [Derived] Abarbanel DN, Seki SM, Davies Y, Marlen N, Benavides JA, Cox K, Nadeau KC, Cox KL. Immunomodulatory effect of vancomycin on Treg in pediatric inflammatory bowel disease and primary sclerosing cholangitis. J Clin Immunol. 2013 Feb;33(2):397-406. doi: 10.1007/s10875-012-9801-1. Epub 2012 Oct 9. PMID 23054338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by the Physician and research team at Lucille Packard and Stanford Hospital and Clinics from 2007 - 2010. The first participant was enrolled in November 2008, and the last participant was enrolled in October 2010.
Pre-assignment Details: 11 PSC patients whose consent to participate was obtained did not participate in the Study.
Groups:
- Oral Vancomycin-Biliary Atresia: Vancomycin: Oral 50mg/Kg per day for three months. Initially 10 infants with Biliary Atresia (BA) were planned for this study to determine if there was clinical response to oral vancomycin.
- Oral Vancomycin/ Primary Sclerosing Cholangitis: Vancomycin: Oral 50mg/Kg per day up to maximum of 1500 mg a day for three months. Initially 10 children with Primary Sclerosing Cholangitis (PSC) were planned for this study to determine if there was clinical response to oral vancomycin.
Period: Overall Study
Arm/Group | Oral Vancomycin-Biliary Atresia | Oral Vancomycin/ Primary Sclerosing Cholangitis
Started | 10 | 11
Completed | 10 | 9
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Based on the annual progress report sent dated 10/04/2010, all patients completed the study as planned except 2 children with PSC- 1 was non-compliant and the other had severe UC requiring Remicade which resulted in removal from Vancomycin study.
Groups:
- Oral Vancomycin-BIliary Atresia: Enrolled- 10, Participated - 10,Completed - 10 (Based on Annual Progress Report in Oct 2010)
- Oral Vancomycin - PSC: Enrolled- 11, Participated - 10 ,Completed - 9 (Based on Annual Progress Report in Oct 2010)
- Total: Total of all reporting groups
Arm/Group | Oral Vancomycin-BIliary Atresia | Oral Vancomycin - PSC | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Customized [Number; unit: participants]
  1-3 months | 10 | 0 | 10
  2-4 years | 0 | 3 | 3
  9-11 years | 0 | 2 | 2
  12-16 years | 0 | 6 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5 | 10 | 15
  Hispanic | 3 | 1 | 4
  African American | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Determine the Benefit of Oral Vancomycin Therapy for Primary Sclerosing Cholangitis and Biliary Atresia
Description: Determine the benefit of oral vancomycin therapy for Primary Sclerosing Cholangitis and Biliary Atresia through improvement of Liver function tests (LFTs) within 3 months of initiating therapy. In addition for PSC, we looked at 25% reduction of abnormal ALT & GGT, reduction in biliary strictures and beading, and reduction of inflammation in liver biopsies and colon biopsies.
Time Frame: Within 3 months of therapy
Population: Ten BA participants had surgery (Kasai portoenterostomyprocedure) at 1 week before starting the Vancomycin so we could not determine if they benefited from the therapy. On oral vancomycin, 9 PSC patients had improvement of LFTs, 8 had improvement of liver biopsies and/or MRI, and colon biopsies,and 1 pt. refused to have these additional studies.
Measure: Number; unit: participants
Groups:
- Liver Blood Test: BA -10/10 , PSC - 9/9 - All had improvement on Vancomycin therapy.
- MRI / MRCP: BA-N/A, PSC - 7/7 showed improvement on Vancomycin therapy.
- Liver Biopsy: BA - N/A , PSC - 4/4 who had Liver biopsies showed improvement on Vancomycin therapy.
- Colon Biopsies: BA - N/A , PSC - 8/8- who had colonoscopies with colon biopsies showed improvement on Vancomycin therapy.
- Liver Biopsy and/or MRI: BA-N/A , PSC- 8/9 participants showed improvement of liver biopsies and/or MRI on Vancomycin.
Arm/Group | Liver Blood Test | MRI / MRCP | Liver Biopsy | Colon Biopsies | Liver Biopsy and/or MRI
Number analyzed (Participants) | 19 | 7 | 4 | 8 | 9
participants
  "BA (n=10,0,0,0,0)" | 10 | 0 | 0 | 0 | 0
  "PSC (n=9,7,4,8,8)" | 9 | 7 | 4 | 8 | 8

ADVERSE EVENTS:
Time Frame: 2 years
Description: There were no adverse experiences for any body system for any participants related to the study that resulted in patients being taken off the study. Since Oral Vancomycin is poorly absorbed, no serious adverse events were anticipated for this study.
Groups:
- BA/PSC -Oral Vancomycin: Oral Vancomycin is commercially available (Vancocin, ViroPharma Inc.) for treatment of gastrointestinal infection such as, Clostridium difficile infection. In fact, our published observation of using oral vancomycin in treating PSC was an incidental finding to our treatment for Cl. Difficile gastrointestinal infection in a child with PSC (J Pediatr Gastroenterol Nutr 27:580-3, 1998). Since oral vancomycin is poorly absorbed, no serious adverse events were anticipated in this study.
Arm/Group | BA/PSC -Oral Vancomycin
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BA/PSC -Oral Vancomycin (N=21)
Non-malignant Spinal Cord Tumor (Nervous system disorders) | 1 (1) — One subject did have a Serious Adverse Event (SAE) that was not related to the study medication or any study procedure. The SAE was for a Non-Malignant Spinal Cord Tumor. This was identified on February 3,2011 and removed on February 18,2011.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes